CLINICAL TRIAL: NCT07007312
Title: Phase 3 Randomized, Double-blind, Placebo-controlled Studies Assessing Ziftomenib in Combination With Either Standard of Care Nonintensive (Venetoclax+Azacitidine) or Intensive (7+3) Therapy in Patients With Untreated NPM1 Mutated or KMT2A Rearranged Acute Myeloid Leukemia
Brief Title: Studies to Assess Ziftomenib in Combination With Ven+Aza or 7+3 in Patients With Untreated NPM1-m or KMT2A-r AML
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KO-MEN-017; 2025-521314-25-00 (EU CTIS Number)
Expanded Access: NCT05738538 (Available)
Record Dates: First submitted 2025-05-16; First posted 2025-06-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: AML; Hematological malignancy; KMT2A; NPM1; Menin; Acute Leukemia; Leukemia; Acute Myeloid Leukemia; Newly diagnosed AML; Newly diagnosed KMT2A-r AML; Newly diagnosed NPM1m AML; Untreated AML; Untreated NPM1m AML; Untreated KMT2A-r AML; MLL
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Hematologic Neoplasms; Leukemia | interventions — venetoclax; Azacitidine; Daunorubicin; Cytarabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Nonintensive Therapy Study, Arm A (Experimental): Ziftomenib in combination with venetoclax+azacitidine
  Interventions: Drug: Ziftomenib; Drug: Venetoclax; Drug: Azacitidine (AZA)
- Nonintensive Therapy Study, Arm B (Placebo Comparator): Placebo in combination with venetoclax+azacitidine
  Interventions: Drug: Placebo; Drug: Venetoclax; Drug: Azacitidine (AZA)
- Intensive Therapy Study, Arm A (Experimental): Ziftomenib+cytarabine+daunorubicin (induction), ziftomenib+cytarabine (consolidation), ziftomenib (maintenance)
  Interventions: Drug: Ziftomenib; Drug: Daunorubicin; Drug: Cytarabine (Ara-C)
- Intensive Therapy Study, Arm B (Experimental): Ziftomenib+cytarabine+daunorubicin (induction), ziftomenib+cytarabine (consolidation), placebo (maintenance)
  Interventions: Drug: Ziftomenib; Drug: Placebo; Drug: Daunorubicin; Drug: Cytarabine (Ara-C)
- Intensive Therapy Study, Arm C (Placebo Comparator): Placebo+cytarabine+daunorubicin (induction), placebo+cytarabine (consolidation), placebo (maintenance)
  Interventions: Drug: Placebo; Drug: Daunorubicin; Drug: Cytarabine (Ara-C)

INTERVENTIONS:
Drug: Ziftomenib — Oral administration
  Other Names: KO-539
  Arms: Intensive Therapy Study, Arm A; Intensive Therapy Study, Arm B; Nonintensive Therapy Study, Arm A
Drug: Placebo — Oral administration
  Arms: Intensive Therapy Study, Arm B; Intensive Therapy Study, Arm C; Nonintensive Therapy Study, Arm B
Drug: Venetoclax — Oral administration
  Other Names: Venclexta; Venclyxto
  Arms: Nonintensive Therapy Study, Arm A; Nonintensive Therapy Study, Arm B
Drug: Azacitidine (AZA) — Intravenous or subcutaneous administration
  Other Names: Vidaza; Azadine
  Arms: Nonintensive Therapy Study, Arm A; Nonintensive Therapy Study, Arm B
Drug: Daunorubicin — Intravenous administration
  Other Names: Cerubidine; daunomycin
  Arms: Intensive Therapy Study, Arm A; Intensive Therapy Study, Arm B; Intensive Therapy Study, Arm C
Drug: Cytarabine (Ara-C) — Intravenous administration
  Other Names: cytosine arabinoside (ara-C); Cytosar-U; Tarabine PFS
  Arms: Intensive Therapy Study, Arm A; Intensive Therapy Study, Arm B; Intensive Therapy Study, Arm C

SUMMARY:
Ziftomenib is an investigational drug in development for the treatment of patients with acute myeloid leukemia (AML) with eligible genetic alterations. Ziftomenib is a type of therapy known to target the menin pathway in cancer cells.

This protocol has 2 separate studies that will investigate the benefits and risks of adding ziftomenib to standard-of-care (SOC) AML treatments in patients with certain genetic mutations who have not received any treatment for their AML. In the first study, the Nonintensive Therapy Study, older patients or those with serious medical problems will receive the SOC therapies venetoclax (ven) and azacitidine (aza), plus either ziftomenib or a placebo. In the second study, the Intensive Therapy Study, medically fit patients will receive (a) the SOC therapies cytarabine and daunorubicin, plus either ziftomenib or a placebo during a first treatment phase called induction, (b) cytarabine plus either ziftomenib or a placebo during a second treatment phase called consolidation, and (c) ziftomenib or a placebo during a third treatment phase called maintenance.

The physician will determine which study is the appropriate treatment for the patient, but neither the patient nor their physician will know whether the patient has been assigned to receive ziftomenib or a placebo. This design is called "double-blinded".

DETAILED DESCRIPTION:
This protocol encompasses two phase 3, randomized, double-blind, placebo-controlled clinical studies to assess the efficacy, safety, and tolerability of ziftomenib in combination with: (a) the standard of care (SOC) nonintensive regimen (venetoclax [ven]+azacitidine [aza]) in untreated adults with nucleophosmin 1 mutated (NPM1-m) acute myeloid leukemia (AML); or (b) the SOC intensive regimen (cytarabine+daunorubicin induction, referred to here as 7+3, and cytarabine consolidation) in untreated adults with NPM1-m or lysine[K]-specific methyltransferase 2A rearranged (KMT2A-r) AML, as well as a maintenance phase.

Nonintensive Therapy Study (Ven+Aza)

Eligible NPM1-m patients will be enrolled and randomized to receive:

* Arm A: Ziftomenib in combination with ven+aza or
* Arm B: Placebo in combination with ven+aza.

Patients will be randomized to treatment arms in a double-blind manner.

Intensive Therapy Study (Cytarabine+Daunorubicin)

Eligible NPM1-m or KMT2A-r patients will be enrolled and randomized to 1 of the following treatment arms:

* Arm A: Ziftomenib+7+3 (induction), ziftomenib+cytarabine (consolidation), ziftomenib (maintenance) or
* Arm B: Ziftomenib+7+3 (induction), ziftomenib+cytarabine (consolidation), placebo (maintenance) or
* Arm C: Placebo+7+3 (induction), placebo+cytarabine (consolidation), placebo (maintenance).

Patients will be randomized to treatment arms in a double-blind manner.

ELIGIBILITY:
Key Inclusion Criteria:

The following criteria apply to both the Nonintensive Therapy Study and the Intensive Therapy Study unless otherwise noted:

* Age ≥18 years at time of signing the informed consent form.
* Diagnosis of AML per the 2022 WHO Classification of Hematolymphoid Tumors (5th Edition).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Adequate liver and kidney function according to protocol requirements.
* A female of childbearing potential must agree to use adequate contraception from the time of screening through 180 days following the last dose of study intervention. A male with a female partner of childbearing potential must agree to use abstinence or adequate contraception from the time of screening through 90 days following the last dose of study intervention.
* NONINTENSIVE THERAPY STUDY ONLY (VEN+AZA):

  1. Documented NPM1-m.
  2. Patients considered ineligible for Intensive Therapy defined by the following:

     * i. Age ≥75, OR
     * ii. Age <75 with an ECOG performance status of 2 or cardiac, renal, or kidney impairment per protocol criteria.
* INTENSIVE THERAPY STUDY ONLY (7+3):

  1. Documented NPM1-m or KMT2A-r (KMT2A-r patients with a partial tandem duplication are not eligible).
  2. Documented FLT3 wild-type or ITD ratio <0.05 OR ineligible to receive FLT3-targeted therapy (medically ineligible or mutation in which FLT3 inhibition is not SOC). Lack of access to an FLT3 inhibitor is not considered "ineligible" for FLT3-targeted therapy.
  3. Ejection fraction of ≥50%.
  4. Fit for Intensive Therapy per Investigator opinion.

Key Exclusion Criteria:

* Prior therapy for AML (except hydroxyurea or leukapheresis for WBC control).
* Diagnosis of acute promyelocytic leukemia (APL), blast phase chronic myeloid leukemia, or isolated myeloid sarcoma.
* Known history of BCR-ABL mutation.
* History of other active concurrent malignancies prior to study entry except:

  1. Basal cell skin cancer or localized squamous cell cancer of the skin
  2. Previous malignancy confined and locally resected (or treated with other modalities) with curative intent
  3. Prostate or breast cancer receiving adjuvant hormonal therapy.
* Active central nervous system (CNS) involvement by AML.
* Clinical signs/symptoms of leukostasis or white blood cells (WBC) >25×10^9/L prior to start of ziftomenib/placebo. Note: Hydroxyurea and/or leukapheresis are permitted to meet this criterion.
* Known uncontrolled HIV infection or known active hepatitis B virus, hepatitis C virus infection, or other uncontrolled infection.
* Uncontrolled intercurrent illness including but not limited to, cardiac illness as defined in the protocol.
* Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2031-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Nonintensive Therapy Study: (Primary Endpoint for all countries): Overall survival (OS) | Defined as the time from randomization to date of death from any cause, assessed up to 36 months after last patient inclusion
  OS
Nonintensive Therapy Study: (Dual Primary Endpoint for US & US reference countries only): Complete remission (CR) | Assessed up to 36 months after last patient inclusion
  CR rate per European Leukemia Network (ELN) 2022 criteria per Investigator assessment
Intensive Therapy Study: (Primary Endpoint for all countries): Event-free survival (EFS) | Defined as the time from randomization to treatment failure, hematologic relapse following CR, or death from any cause, whichever comes first, assessed up to 36 months after last patient inclusion
  EFS
Intensive Therapy Study: (Dual Primary Endpoint for US & US reference countries only): Complete remission (CR) with bone marrow (BM) measurable residual disease (MRD) negativity in NPM1-m patients | Assessed up to 36 months after last patient inclusion
  CR rate per ELN 2022 criteria per Investigator assessment with central BM MRD negativity

SECONDARY OUTCOMES:
Nonintensive Therapy Study: (EU & EU reference countries only): Complete remission (CR) | Up to 36 months after last patient inclusion
  CR rate per ELN 2022 criteria per Investigator assessment
Nonintensive Therapy Study: Bone marrow (BM) measurable residual disease (MRD) negativity | Up to 36 months after last patient inclusion
  Central BM MRD negativity rate
Nonintensive Therapy Study: Complete remission (CR) + complete remission with partial hematologic recovery (CRh) | Up to 36 months after last patient inclusion
  CR + CRh rate per ELN 2022 criteria per Investigator assessment
Nonintensive Therapy Study: Descriptive statistics of Adverse Events (AEs) | From start of treatment to 28 days from last dose of ziftomenib or placebo
  Assessed by NCI-CTCAE v5.0
Nonintensive Therapy Study: Area under the concentration-time curve (AUC) of ziftomenib and venetoclax | During treatment for up to 36 months after last patient inclusion
  To characterize the AUC of ziftomenib and venetoclax
Nonintensive Therapy Study: Trough concentration (Ctrough) of ziftomenib and venetoclax | During treatment for up to 36 months after last patient inclusion
  To characterize the Ctrough of ziftomenib and venetoclax
Nonintensive Therapy Study: Health-related patient-reported outcomes (PRO) assessments | Up to 36 months after last patient inclusion
  Health-related quality of life (HRQoL) was evaluated by EORTC QLQ-C30 global health status/quality of life composite scale in all randomized participants. The QLQ-C30 is a cancer-specific, self-administered questionnaire that contains 30 questions, covering global, functional, and symptom scales. Scores range from 0 to 100. Higher scores on global and functional scales indicated better quality of life (QoL), while higher scores on the symptom scales indicated declining QoL.
Intensive Therapy Study: (EU & EU reference countries only): Complete remission (CR) with bone marrow (BM) measurable residual disease (MRD) negativity in NPM1-m patients | Up to 36 months after last patient inclusion
  CR rate per ELN 2022 criteria per Investigator assessment with central BM MRD negativity
Intensive Therapy Study: Overall survival (OS) | Defined as the time from randomization to date of death from any cause, up to 36 months after last patient inclusion
  OS
Intensive Therapy Study: Descriptive statistics of Adverse Events (AEs) | From start of treatment to 28 days from last dose of ziftomenib or placebo
  Assessed by NCI-CTCAE v5.0
Intensive Therapy Study: Health-related patient-reported outcomes (PRO) assessments | Up to 36 months after last patient inclusion
  Health-related quality of life (HRQoL) was evaluated by EORTC QLQ-C30 global health status/quality of life composite scale in all randomized participants. The QLQ-C30 is a cancer-specific, self-administered questionnaire that contains 30 questions, covering global, functional, and symptom scales. Scores range from 0 to 100. Higher scores on global and functional scales indicated better quality of life (QoL), while higher scores on the symptom scales indicated declining QoL.
Intensive Therapy Study: Area under the concentration-time curve (AUC) of ziftomenib | During treatment for up to 36 months after last patient inclusion
  To characterize the AUC of ziftomenib
Intensive Therapy Study: Trough concentration (Ctrough) of ziftomenib | During treatment for up to 36 months after last patient inclusion
  To characterize the Ctrough of ziftomenib

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - University of California, San Diego, La Jolla, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Kentucky, Lexington, Kentucky
  - Wayne State University School of Medicine, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Rutgers Biomedical and Health Sciences, New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Willamette Valley Cancer Institute, Eugene, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology-Presbyterian Cancer Center, Dallas, Texas
  - University of Texas, Houston, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - University of Virginia School of Medicine, Charlottesville, Virginia
  - Virginia Cancer Specialists, Manassas, Virginia

IPD SHARING:
Plan to Share IPD: Undecided